CLINICAL TRIAL: NCT00004757
Title: Phase III Randomized, Placebo-Controlled Study of Acyclovir Oral Suspension for Neonatal Herpes Simplex Virus Infection Limited to the Skin, Eyes, and Mouth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11687; NIAID-558609
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-01

CONDITIONS: Herpes Simplex
Keywords: herpes simplex virus infection; herpesvirus infection; immunologic disorders and infectious disorders; rare disease; viral infection
MeSH Terms: conditions — Herpes Simplex; Herpesviridae Infections; Immune System Diseases; Communicable Diseases; Rare Diseases; Virus Diseases | interventions — Acyclovir

INTERVENTIONS:
Drug: acyclovir

SUMMARY:
OBJECTIVES: I. Determine whether acyclovir (ACV) oral suspension suppresses recurrent skin lesions and improves neurologic outcome in neonates with localized herpes simplex virus type 2 infection when administered for 6 months in a placebo-controlled study.

II. Determine whether the prevention of recurrent skin lesions reduces long-term neurologic morbidity.

III. Determine whether resistant disease develops after oral ACV therapy. IV. Evaluate the natural history of recurrent skin lesions. V. Measure any adverse effects and laboratory abnormalities associated with long-term oral ACV therapy in infants and young children.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by participating institution.

All patients are treated with intravenous acyclovir for 14 days. Patients are then randomly assigned to 1 of 2 treatment groups if the following criteria are met: no systemic disease involvement, documented by negative cerebrospinal fluid exam, brain computerized tomography, and magnetic resonance imaging; and entry criteria continue to be met.

Randomized treatment begins 8 hours after the final dose of intravenous acyclovir. One group is treated with oral acyclovir, while the control group receives an oral placebo.

Treatment continues for 6 months in the absence of unacceptable toxicity, systemic disease, and 2 or more recurrences of skin lesions. Patients are followed at 6 months, then yearly for at least 4 years.

The study duration is estimated to be 4 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Virologically confirmed herpes simplex virus type 2 (HSV-2) with skin lesions localized to the skin, eyes, and mouth
* No central nervous system or disseminated disease Normal cerebrospinal fluid WBC less than 20 Protein less than 90 mg/dL
* Normal brain computerized tomography or magnetic resonance imaging (MRI) MRI if feasible
* No HSV-1

--Patient Characteristics--

* Age: Under 29 days
* Renal: Creatinine no greater than 1.5 mg/dL
* Other: Birth weight at least 1200 g
* Gestational age greater than 32 weeks
* No breast feeding if mother on acyclovir

Ages: 0 Years to 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1992-08

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Whitley, Study Chair — National Institute of Allergy and Infectious Diseases (NIAID)